CLINICAL TRIAL: NCT03756025
Title: Atraumatic Restorative Treatment (ART) in Early Childhood Caries in Brazilian Babies: a Longitudinal Randomized Clinical Trial
Brief Title: Atraumatic Restorative Treatment (ART) in Early Childhood Caries (ECC)
Acronym: ART-ECC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Daniel Demétrio Faustino da Silva, Principal Investigator, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ART-ECC
Record Dates: First submitted 2018-11-21; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Early Childhood Caries
Keywords: Early Childhood Caries; Atraumatic Restorative Treatment; Glass Ionomer Cement; Deciduous Tooth; Odontopediatrics
MeSH Terms: interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Intervention Model Description: The study is characterized by longitudinal follow-up of a randomized, double-blind, split-mouth-type clinical trial performed in babies affected by early childhood caries
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each evaluation was performed by a different blind examiner for the type of GIC used in ART Patients did not know what material was being used on their teeth.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitro Molar® (DFL, Rio de Janeiro, Brazil) (Experimental): ART restorations of a face with one of the two high-viscosity conventional glass ionomer cements-Vitro Molar® (DFL, Rio de Janeiro, Brazil).
  Interventions: Procedure: Atraumatic Restorative Treatment (ART)
- Ketac Molar Easy Mix® (3M ESPE, St Paul, MN, USA). (Active Comparator): ART restorations of a face with one of the two high-viscosity conventional glass ionomer cements-Ketac Molar Easy Mix® (3M ESPE, St Paul, MN, USA).
  Interventions: Procedure: Atraumatic Restorative Treatment (ART)

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment (ART) — The atraumatic restorations were performed in the dental office by a single operator trained in the ART Technique [20], who received the restorative material already prepared by a trained auxiliary, ensuring blinding of the study. The restorative procedure performed in relative isolation and without the use of anesthesia consisted of removal of the carious tissue using hand instrument excavators and dentin spoons, with subsequent conditioning of the cavity with a polyacrylic acid solution at 11.5% (DFL) applied with a microbrush for 10 seconds. Immediately after, the cavity was washed and dried with cotton balls. In this step, according to the randomization, the respective GIC was inserted and subsequent digital compression was performed for 30 seconds. After occlusal adjustment, the ARTs were protected with finish gloss Alfa Bond® (DFL).
  Other Names: ART

SUMMARY:
Considering the severity and high prevalence of ECC, as well as the importance of early intervention and approach, the Atraumatic Restorative Treatment program, because of its advantages, consists of an important treatment alternative. However, only a few studies assess ART in babies affected by ECC. For this practice to be accepted as safe, scientific evidence must be built through longitudinal studies to evaluate ART performance and to this end, the present study is justified. Therefore, the aim of this research was to evaluate the effectiveness of Atraumatic Restorative Treatment performed in babies suffering from ECC after a 4-year period and compare the clinical performance of Atraumatic Restorations performed with two different glass ionomer cements. The investigator's hypothesis is that there is no difference in the clinical performance of ARTs performed with the different GICs.

The study is characterized by longitudinal follow-up of a randomized, double-blind, split-mouth-type clinical trial performed in babies affected by early childhood caries. The subjects were children of both sexes, aged between 18 and 36 months, with at least one deciduous molar in each of the different dental quadrants, presenting active cavitated lesions of shallow or medium depth, involving only the occlusal surface. The initial convenience sample consisted of 100 deciduous molars of 25 children attending Bebê Clínica of the School of Dentistry of the Federal University of Rio Grande do Sul-FO / UFRGS, Porto Alegre-RS, Brazil;

DETAILED DESCRIPTION:
The study is characterized by longitudinal follow-up of a randomized, double-blind, split-mouth-type clinical trial performed in babies affected by early childhood caries. The subjects were children of both sexes, aged between 18 and 36 months, with at least one deciduous molar in each of the different dental quadrants, presenting active cavitated lesions of shallow or medium depth, involving only the occlusal surface. The initial convenience sample consisted of 100 deciduous molars of 25 children attending Bebê Clínica of the School of Dentistry of the Federal University of Rio Grande do Sul-FO / UFRGS, Porto Alegre-RS, Brazil; this number being based on similar studies published in the literature [27, 28, 29]. The power of the sample was calculated using the PEPI program, version 4 (Computer Programs for Epidemiologists), for a significance level of 5%. Considering that the average success percentage in two years of ART on primary teeth facings was 88%, and the worst result found was 67% [30], the power obtained was of 70.1%.

All children in the study were enrolled in the oral health promotion program for babies, in which mothers accompanied by their children individually received information and guidance on food intake, breastfeeding, and oral hygiene. In addition to the guidance that was reinforced at each visit, children received topical application of fluoride by brushing with acidulated phosphate fluoride gel in four applications with intervals of one week, considering that all had active cavities [31].

The clinical trial was performed through the experimental split-mouth model, in which the 25 selected children had their teeth distributed randomly through a random number table, receiving ART restorations of a face with one of the two high-viscosity conventional glass ionomer cements studied: Vitro Molar® (DFL, Rio de Janeiro, Brazil) and Ketac Molar Easy Mix® (3M ESPE, St Paul, MN, USA). The atraumatic restorations were performed in the dental office by a single operator trained in the ART Technique [20], who received the restorative material already prepared by a trained auxiliary, ensuring blinding of the study. The restorative procedure performed in relative isolation and without the use of anesthesia consisted of removal of the carious tissue using hand instrument excavators and dentin spoons, with subsequent conditioning of the cavity with a polyacrylic acid solution at 11.5% (DFL) applied with a microbrush for 10 seconds. Immediately after, the cavity was washed and dried with cotton balls. In this step, according to the randomization, the respective GIC was inserted and subsequent digital compression was performed for 30 seconds. After occlusal adjustment, the ARTs were protected with finish gloss Alfa Bond® (DFL).

Clinical assessments were carried out in three stages: after 1, 2 and 4 years. For this, the oral health status of the children was assessed by the presence of visible plaque and caries activity, and the quality of ART restorations by the ART criterion [20]. In the exams at 4 years, an additional assessment was done by means of the modified United States Public Health Service (USPHS) criteria [32] and the Visible Plaque Index-VPI and Gingival Bleeding Index-GBI [33]. Each evaluation was performed by a different blind examiner for the type of GIC used in ART and calibrated with the respective intra-examiner correlation coefficients: 1 year (ART Criterion: Kappa=0.81), 2 years (ART Criterion: Kappa=0.83), and 4 years (ART Criterion: Kappa=0.86; Modified USPHS Criteria: Kappa average=0.73; VPI: Kappa=0.79; caries activity: Kappa=1.0).

For the analysis of the general clinical performance of ART, through the success rate among the different GICs, the chi-square test was applied. In addition, the Mann-Whitney test was used to compare each individual clinical criterion between the materials (retention and anatomical shape, integrity and marginal discoloration, color of material, surface roughness and secondary caries), with all tests at the level of significance of 5% (p <0.05). The Visible Plaque Index (VPI) and Gingival Bleeding Index (GBI), as well as caries activity were expressed through frequencies distribution.

Database construction and analysis, and interpretation of results were obtained by using the Statistical Package for the Social Sciences (SPSS), version 19.0.

ELIGIBILITY:
Inclusion Criteria:

* presence of active carious cavitated lesions;
* least one deciduous molar in each of the different dental quadrants;
* caries of shallow or medium depth, involving only the occlusal surface.

Exclusion Criteria:

* Children who do not allow clinical procedures to be performed.

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2008-12-31 (Actual); Study Completion 2009-06-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance scale of restaruations through the ART(Atraumatic Restorative Treatment ) criterion. | Through study completion, an average of 1 year
  Success: Codes 0(Present, satisfactory), 1(Present, slight deficiency at cavity margin of less than 0.5 mm) and 7(Not present, other restorative treatment performed)
Clinical performance scale of restaruations through the ART(Atraumatic Restorative Treatment ) criterion. | Through study completion, an average of 1 year
  Failure: Codes 2(Present, deficiency at cavity margin of 0.5 mm or more), 3(Present, fracture in restoration), 4(Present, fracture in tooth), and 8(Not present, tooth is not present)

SECONDARY OUTCOMES:
Clinical performance scale of restaruations through the USPHS(United States Public Health Service ) criteria. | Through study completion, an average of 1 year
  Success: Codes A=Alfa (Restoration is intact and fully retained) and B=Bravo (Restoration is partially retained with some portion of the restoration still intact)
Clinical performance scale of restaruations through the USPHS(United States Public Health Service ) criteria. | Through study completion, an average of 1 year
  Failure: Codes C(Restoration is completely missing)

CONTACTS AND LOCATIONS:
Locations (1):
- Nossa Senhora da Conceição Hospital, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faustino-Silva DD, Figueiredo MC. Atraumatic restorative treatment-ART in early childhood caries in babies: 4 years of randomized clinical trial. Clin Oral Investig. 2019 Oct;23(10):3721-3729. doi: 10.1007/s00784-019-02800-8. Epub 2019 Jan 21. PMID 30666480